CLINICAL TRIAL: NCT05354908
Title: Surgical Research in Colombia Part 1: Scientific and Academic Productivity of the Colombian Research Groups in Surgery
Brief Title: Surgical Research in Colombia Part 1
Status: Completed | Type: Observational
Sponsor: Ivan David Lozada-Martinez (Other)
Responsible Party: Sponsor-Investigator, Ivan David Lozada-Martinez, Principal Investigator, Colombian Surgery Association
Organization: Colombian Surgery Association (Other)
Other Study IDs: 00001
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Academic Productivity; Research Productivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colombian research groups in surgery: Colombian research groups in surgery
  Interventions: Other: scientific and academic productivity

INTERVENTIONS:
Other: scientific and academic productivity — Number and quartile of scientific products generated by the group

SUMMARY:
Global surgery has become the undisputed starting point for addressing a myriad of problems in surgery today. Therefore, it is necessary to constantly evaluate the scientific productivity in surgery, its behavior, validity and impact. In Latin America, specifically in Colombia, there are no studies that have analyzed this production. A retrospective cross-sectional bibliometric study was carried out, in which the Colombian Ministry of Science database was consulted with the validated results up to July 2021. In the search section for research groups, the keyword "Surgery" was used, and all associated Groups in Latin America and the Caribbean(platform where the information of the research groups can be found) and their registered products were reviewed

ELIGIBILITY:
Inclusion Criteria:

* Research groups with a main or secondary line of research in general or subspecialty surgery, registered in the base of the Colombian Ministry of Science

Exclusion Criteria:

* Research groups with other lines of research in the surgical sciences

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Research groups recognized and/or categorized by the Colombian Ministry of Science
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Number of articles published in journals indexed in SJR, Scopus or JCR | 1 year
  Frequency of articles of any type published in journals indexed in the Scimago Journal Rank, Scopus and Journal Citation Report databases
Quartile of journals in which the articles registered in the database were published | 1 year
  Quartile of the article according to the quartile of the journal in which it was published

SECONDARY OUTCOMES:
Graduate students' theses supervised by the research group | 1 year
  Number of theses supervised by the research group
Type of graduate students' theses supervised by the research group | 1 year
  Category of registered graduate thesis by the research group
Frequency of attendances and presentations at scientific events | 1 year
  Number of attendances and presentations in scientific events in medicine
Type of participation in scientific events in medicine | 1 year
  Category of participation of the scientific event in medicine
Research projects registered by the research group | 1 year
  Number research project registered and declared up to the date of the study
Type of research projects registered by the research group | 1 year
  Category of research project registered and declared up to the date of the study
Book chapters published by the research group to date | 1 year
  Frequency of publication of book chapters by the research group
Books published by the research group to date | 1 year
  Frequency of publication of book by the research group

CONTACTS AND LOCATIONS:
Locations (1):
- Colombian Ministry of Science Database, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
This data is available to the public